CLINICAL TRIAL: NCT03364283
Title: The Effects of Sitting Position on the Outcome During Surgery on Posterior Cranial Fossa and Pineal Region
Brief Title: Sitting Versus Horizontal Position on Craniotomies
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Burdenko Neurosurgery Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2015H0035
Record Dates: First submitted 2017-10-04; First posted 2017-12-06 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Craniotomy; Brain Tumor
Keywords: Posterior fossa; Pineal region
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sitting Position: Sitting and semi-sitting
  Interventions: Procedure: Surgical position
- Horizontal Position: Prone, lateral and park bench.

INTERVENTIONS:
Procedure: Surgical position
  Groups: Sitting Position

SUMMARY:
The main objectives of this study are comparison of the incidence of intraoperative air embolism and the extent of blood loss in patients undergoing posterior cranial fossa (PCF) and pineal region (PR) surgeries in sitting and horizontal position. Additionally, the overall treatment outcome, neurological functional outcome, degree of tumor removal, clinical course in the postoperative period, and the patient satisfaction will be compared between the groups.

DETAILED DESCRIPTION:
This was a prospective observational study to assess the effects of patient positioning during craniotomies on surgical outcomes. Patients were distributed into 2 major groups based on the surgical position: sitting and horizontal. Each group was further divided into subgroups based on the type and location of the lesion. To achieve the study goals, comparison of the 2 approaches in equivalent patient groups was performed, including comparable demographics, diagnoses, topographic location of the lesions, anesthetic approaches, and surgical experience.

The operating surgeons decided patient positioning based on clinical judgment. Type of anesthesia was defined by the anesthesiologist in charge of the patient however, it was maximally standardized for both sites. All the surgeries were performed by neurosurgeons with sufficient experience of sitting craniotomies.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 - 75 years old undergoing open posterior cranial fossa and pineal region surgery and diagnosed with space-occupying or vascular lesions willing consent to participate in the study.

Exclusion Criteria:

* Significant cardio-vascular comorbid conditions (cardiac insufficiency, recent infarction, advanced arterial hypertension)
* Advanced chronic respiratory comorbid conditions
* Uncorrected hypovolemia, anemia, hypoalbuminemia
* De-compensated acid base and electrolyte disorders
* Anticoagulated patients and patients with coagulation disorders, deep venous thrombosis (history of deep vein thrombosis or clinically established)
* Preoperative evidence of spinal or peripheral nerve dysfunction that may interfere with patient positioning.
* Cervical myelopathy
* Cervical spine disorders (atlanto-occipital arthritis, previous fractures etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective craniotomies on posterior cranial fossa or pineal region were identified on each site before surgery. Patients were asked to be part of the study explaining that no intervention was necessary besides a phone call performed by the research team 3 months after their surgery.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative air embolism | Time of surgery (From surgical wound incision time until wound closure)
  Measured intraoperatively with transesophageal echocardiogram and/or PETCO2 levels

SECONDARY OUTCOMES:
Degree of tumor removal | End of surgery (closure) - Postoperative evaluation by surgeon and/or postoperative imaging performed up to 48 hours after end of surgery
  Indicated by surgeon description and/or postoperative imaging
Neurological function | End of surgery (closure) - Discharge from the hospital or up to 3 months after end of surgery, whichever came first.
  Compared sensory-motor function, cranial nerve function and Glasgow scale before and after surgery.
Patient satisfaction | End of surgery (closure) - 3 months after surgery
  Collected on phone script during follow-up phone call

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Bergese, MD, Principal Investigator — Ohio State University

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication

REFERENCES:
- [Derived] Mavarez-Martinez A, Israelyan LA, Soghomonyan S, Fiorda-Diaz J, Sandhu G, Shimansky VN, Ammirati M, Palettas M, Lubnin AY, Bergese SD. The Effects of Patient Positioning on the Outcome During Posterior Cranial Fossa and Pineal Region Surgery. Front Surg. 2020 Mar 13;7:9. doi: 10.3389/fsurg.2020.00009. eCollection 2020. PMID 32232048